CLINICAL TRIAL: NCT00004690
Title: Phase III Study of Monolaurin Cream Therapy for Patients With Congenital Ichthyosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cellegy Pharmaceuticals (Industry)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13316; CELLEGY-FDR001278
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Ichthyosis
Keywords: dermatologic disorders; ichthyosis; rare disease
MeSH Terms: conditions — Ichthyosis; Skin Diseases; Rare Diseases

INTERVENTIONS:
Drug: monolaurin cream

SUMMARY:
OBJECTIVES: I. Compare the safety and efficacy of monolaurin cream versus a placebo vehicle cream in suppressing the signs of nonbullous congenital ichthyosiform erythroderma.

II. Assess the incidence of posttreatment rebound or recrudescence in patients with congenital ichthyosis.

III. Evaluate the long term safety of monolaurin cream with whole body application in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a three month, randomized, double blind, placebo controlled study followed by a nine month, open label, rollover study.

Patients are treated either with a placebo vehicle cream or the study cream, monolaurin (15% glyceryl monolaurate), for 3 months followed by a four week break. Medications are applied uniformly twice daily (morning and at least 1 hour before bedtime). After this blinded portion of the study, all patients are administered monolaurin cream for 9 months.

Patients are followed for 4 weeks after the last cream application.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Nonbullous congenital ichthyosiform erythroderma (chronic, multifactorial, hyperkeratotic, inflammatory skin disease) Clinical criteria includes: - generalized involvement with no flexural sparing - congenital onset usually as collodion baby (i.e., a taut, shiny encasement which is shed postnatally revealing underlying erythroderma and generalized ichthyosis) - scales should be fine, whitish, and rather loose except on the lower legs where the scales may be large, platelike, and dark - if severely effected: intense erythema is present; overt ectropion may be present; cicatricial alopecia may be present; and secondary nail dystrophies with thickening of nail plate and ridging may be present
* Phenotypically consistent with diagnostic grading photos
* Grade of at least 3 for scaling on four treatment sites

--Prior/Concurrent Therapy--

* Biologic therapy: Not specified
* Chemotherapy: Not specified
* Endocrine therapy: At least 4 weeks since prior corticosteroids No concurrent corticosteroids
* Radiotherapy: Not specified
* Surgery: Not specified
* Other: At least 4 weeks since any prior investigational medications At least 4 weeks since any prior systemic therapy, such as hypolipidemics or retinoids Nonglycerin emollients allowed up to 1 week prior to study At least 4 weeks since any other topical therapy including humectants such as urea, alpha hydroxy or alpha ketoacid preparations and retinoids No concurrent topical therapy No concurrent investigational medications

--Patient Characteristics--

* Age: 18 months and over
* Performance status: Not specified
* Hematopoietic: No clinically significant laboratory abnormalities
* Hepatic: No clinically significant laboratory abnormalities
* Renal: No clinically significant laboratory abnormalities
* Other: Triglyceride or total cholesterol no greater than 3 times normal Must be in general good health No known hypersensitivity to any component of this study medication Not pregnant or nursing Adequate contraception required of all fertile women

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1996-09; Study Completion 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Carl R. Thornfeldt, Study Chair — Cellegy Pharmaceuticals